CLINICAL TRIAL: NCT03410316
Title: The Netherlands Epidemiology of Obesity Study
Acronym: NEO
Status: Active, not recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, FritsRRosendaal, MD PhD, Leiden University Medical Center
Other Study IDs: P08.109
Record Dates: First submitted 2018-01-10; First posted 2018-01-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: Obesity; Common diseases; Epidemiology; Etiology
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Urine
  * Plasma
  * Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants of the NEO study: Men and women aged 45 oy 65 years, with an oversampling of individuals with a BMI of 27 kg/m2 or higher
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The Netherlands Epidemiology of Obesity (NEO) study is a population-based cohort study in 6671 men and women aged 45 to 65 years, with an oversampling of individuals with a BMI of 27 kg/m2 or higher. The NEO study is designed to investigate pathways that lead to common diseases and conditions.

Men and women aged between 45 and 65 years with a self-reported BMI of 27 kg/m2 or higher living in the greater area of Leiden, the Netherlands, were eligible to participate in the NEO study. Participants were recruited via three recruitment strategies. First, participants were recruited by general practitioners in the area of Leiden, in the West of The Netherlands. Second, participants were recruited through advertisements in local newspapers and through posters distributed in public areas of Leiden and surroundings. Third, participants were recruited via the registries of three municipalities surrounding Leiden (Katwijk, Leiderdorp and Teylingen). Inhabitants of Katwijk and Teylingen aged between 45 and 65 years were invited to participate if they had a self-reported BMI of 27 kg/m2 or higher. All inhabitants aged between 45 and 65 years of Leiderdorp were invited to participate irrespective of their BMI, allowing for a reference distribution of BMI.

Participants were invited to a baseline visit at NEO study centre of the LUMC after an overnight fast. Prior to this study visit, participants collected their urine over 24 h and completed a general questionnaire at home to report demographic, lifestyle and clinical information. The participants were asked to bring all medication they were using to the study visit. At the baseline visit an extensive physical examination was performed, including measurements of anthropometry, blood pressure, both fasting and postprandial blood sampling (30 minutes and 2.5 hours after a liquid mixed meal), ECG, carotid artery IMT, and pulmonary function tests. In random subsets of participants MRI of abdominal fat, brain, knee, heart function, and pulse wave velocity of the aorta was performed, as well as indirect calorimetry, accelerometry combined with continuous heart rate, and total sleep time with actigraphy. Participants are followed via their general practitioners and hospital registries for the incidence of common diseases and mortality.

DETAILED DESCRIPTION:
Hypotheses

1. Overweight and obesity affect major systemic responses, such as inflammation and coagulation that lead to the occurrence of major common diseases.
2. The occurrence of these diseases is related to individual make-up, including genetics and fat type and location, and environment, and the interaction between the various systemic responses, and the (subclinical) disease outcomes.

Primary general objectives of the NEO study

1. To study the pathways that lead to common diseases in overweight and obese individuals.
2. To identify novel determinants of various diseases and conditions in overweight and obese individuals.
3. To study interrelationships between diseases, newly identified determinants with each other and with classical, established risk factors.

Secondary general objectives of the NEO Study

1. To identify novel determinants of various subclinical conditions in overweight and obese individuals.
2. To develop novel methods for determining the risk of various diseases and conditions in asymptomatic overweight and obese individuals, in addition to established prognostic markers.
3. To assess the burden of disease in a population-based cohort of overweight and obese individuals.
4. To investigate the optimal diagnostic method to define overweight and obesity in terms of predicting various diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 45 to 65
* Self-reported BMI of 27kg/m2 or higher
* Subgroup of participants irrespective of their BMI

Exclusion Criteria:

* NA

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women living in the greater area of Leiden (in the West of the Netherlands) were invited by letters sent by general practitioners, and via municipalities and by local advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 6671 (Actual)
Dates: Start 2008-08-04 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of common diseases | Around each 5 years
  e.g. type 2 diabetes (yes/no), cardiovascular diseases (y/n), thrombosis (y/n), chronic kidney disease (y/n), asthma (y/n), chronic obstructive pulmonary disease (y/n), osteoarthritis (y/n), cirrhosis (y/n), depression (y/n)

CONTACTS AND LOCATIONS:
Overall Officials: Frits R Rosendaal, Principal Investigator — Department of Clinical Epidemiology, Leiden University Medical Center; Renée de Mutsert, Study Director — Department of Clinical Epidemiology, Leiden University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
This is a publicly funded observational study, all data are owned by the university and open to researchers after consultation and according to internal procedures

REFERENCES:
- [Background] de Mutsert R, den Heijer M, Rabelink TJ, Smit JW, Romijn JA, Jukema JW, de Roos A, Cobbaert CM, Kloppenburg M, le Cessie S, Middeldorp S, Rosendaal FR. The Netherlands Epidemiology of Obesity (NEO) study: study design and data collection. Eur J Epidemiol. 2013 Jun;28(6):513-23. doi: 10.1007/s10654-013-9801-3. Epub 2013 Apr 11. PMID 23576214
- [Derived] Oosterom-Eijmael MJP, le Cessie S, Slats AM, Hiemstra PS, Thijs W, Lamb HJ, Willems van Dijk K, Rosendaal FR, de Mutsert R. The relation between visceral fat and lung function in the general population is in part mediated by CRP and leptin. Expert Rev Respir Med. 2025 Aug;19(8):887-897. doi: 10.1080/17476348.2025.2502557. Epub 2025 Jun 4. PMID 40468646
- [Derived] Winters-VAN Eekelen E, VAN DER Velde JHPM, Boone SC, Westgate K, Brage S, Lamb HJ, Rosendaal FR, DE Mutsert R. Objectively Measured Physical Activity and Body Fatness: Associations with Total Body Fat, Visceral Fat, and Liver Fat. Med Sci Sports Exerc. 2021 Nov 1;53(11):2309-2317. doi: 10.1249/MSS.0000000000002712. PMID 34081059
- [Derived] van Eekelen E, Beulens JWJ, Geelen A, Schrauwen-Hinderling VB, Lamb H, de Roos A, Rosendaal F, de Mutsert R. Consumption of Alcoholic and Sugar-Sweetened Beverages is Associated with Increased Liver Fat Content in Middle-Aged Men and Women. J Nutr. 2019 Apr 1;149(4):649-658. doi: 10.1093/jn/nxy313. PMID 30949667
- [Derived] van Eekelen E, Geelen A, Alssema M, Lamb HJ, de Roos A, Rosendaal FR, de Mutsert R. Sweet Snacks Are Positively and Fruits and Vegetables Are Negatively Associated with Visceral or Liver Fat Content in Middle-Aged Men and Women. J Nutr. 2019 Feb 1;149(2):304-313. doi: 10.1093/jn/nxy260. PMID 30657914